CLINICAL TRIAL: NCT01901380
Title: Effect of Lactobacillus GG on the Appearance of Functional Gastrointestinal Disorders in Children With Cow's Milk Allergy
Brief Title: Cow's Milk Allergy and Functional Gastrointestinal Disorders
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Other Study IDs: 204/12
Record Dates: First submitted 2013-07-03; First posted 2013-07-17 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Cow's Milk Allergy; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Milk Hypersensitivity; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- extensively hydrolysed casein formula + LGG: children receiving extensively hydrolysed casein formula plus Lactobacillus GG
  Interventions: Dietary Supplement: Extensively hydrolyzed casein formula + LGG
- other formulas: children receiving formulas without supplementation of Lactobacillus GG
  Interventions: Dietary Supplement: Extensively hydrolyzed casein formula + LGG

INTERVENTIONS:
Dietary Supplement: Extensively hydrolyzed casein formula + LGG

SUMMARY:
Cow's milk allergy (CMA) is the most common food allergy in early childhood, with an estimated incidence ranging between 2% and 3% in infants and marginally lower in older children. It has been demonstrated that it could be a risk factor for the development of the functional gastrointestinal disorders in children. Intestinal microflora has been indicated as potential target for the management of CMA and FGDIs through the use of probiotics. Lactobacillus rhamnosus GG (LGG) is the most studied probiotic. Recently, it has been demonstrated that an extensively hydrolyzed casein formula remains hypoallergenic following the addition of LGG, satisfying both the American Academy of Pediatrics guidelines. Lactobacillus GG exerts several benefits when added to an extensively hydrolyzed casein formula (Nutramigen LGG), including decreased severity of atopic dermatitis, improved recovery of intestinal symptoms in infants with CMA-induced allergic colitis, and faster induction of tolerance in infants with CMA. The mechanisms of these effects are multiple and exerted at different levels: epithelium, immune system and enteric nervous system. Studies and meta-analyses showed that LGG increases treatment success in children with functional gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Children (aged from 4 to 6 yrs) with a history of sure diagnosis of cow's milk allergy obtained in the first year of life treated with hypoallergenic formula

Exclusion Criteria:

* Age higher than 12 months,
* concomitant chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal tract,
* suspected eosinophilic esophagitis or eosinophilic enterocolitis,
* suspected food-protein-induced enterocolitis syndrome,
* suspected cow's milk proteins-induced anaphylaxis.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be enrolled from a cohort of about 300 children (aged from 4 to 6 yrs) with a history of sure diagnosis of CMA obtained in the first year of life treated with hypoallergenic formula for at least 6 months and who are already in follow-up at the Department of Pediatrics of University of Naples "Federico II".
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Appearance of functional gastrointestinal disorders | functional gastrointestinal disorders

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy